CLINICAL TRIAL: NCT04798859
Title: Treating Chronic Symptoms of Pediatric Acquired Brain Injury - The Child In Context Intervention Study
Brief Title: The Child in Context Intervention Study
Acronym: CICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: The Research Council of Norway (Other); Oslo University Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Monash University (Other); The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SunnaasRH_CICI226059
Record Dates: First submitted 2021-03-02; First posted 2021-03-15 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2022-11

CONDITIONS: Rehabilitation; Brain Injuries; Brain Injury, Chronic; Brain Diseases; Family; Childhood Brain Tumor; Child Behavior; Parenting
Keywords: Pediatric brain injury; Randomized controlled trial (RCT); School; Family health care needs; Community
MeSH Terms: conditions — Brain Injuries; Brain Injury, Chronic; Brain Diseases; Child Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Independent Outcome Assessor(s) will be blinded to group allocation. Participants will be provided with new IDs in final database, blinding researchers to which group is the intervention group during analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-centered in home rehabilitation (Experimental): Seven individualized meetings with the family (7 sessions whereof most will be videoconferences, with the possibility of 1-2 of the sessions being home visits), one parent group seminar and 4 meetings (three videoconferences and one phone call) with school and local care providers during a period of 4-5 months.
  Based on target outcomes areas noted by children and parents, individual goals will be established (2-5 per family). Strategies to meet goals will be established for each goal, and goal attainment scaling will be used to quantify goal attainment.
  Interventions: Other: Family centered in-home rehabilitation
- Control group (Active Comparator): Usual health care and rehabilitation services provided in the municipality, including school.
  Interventions: Other: Control

INTERVENTIONS:
Other: Family centered in-home rehabilitation — Goal-oriented individualized intervention targeting brain injury related areas noted as challenging by the child and family
  Arms: Family-centered in home rehabilitation
Other: Control — Usual follow-up in the municipality
  Arms: Control group

SUMMARY:
Children with acquired brain injury (ABI) often struggle with complex impairments, including cognitive (such as memory and attention), social, emotional and behavioral challenges. There is a lack of evidence-based knowledge about rehabilitation for children with ABI in the chronic phase. The current study, the CICI Study, is a randomized controlled trial (RCT) directed towards children with ABI and their families in the chronic phase.

The study will be conducted in close collaboration with schools and local health care providers. The CICI Study focuses on the child's and parents' individually identified target outcome areas and rehabilitation goals. The intervention aims to enhance everyday functioning in the home and school environment by attaining rehabilitation goals in areas noted as challenging by the participants. The efficacy of the CICI-intervention will be measured in terms of goal attainment, burden of brain injury related symptoms, parenting self-efficacy, unmet health care needs, as well as several aspects of child, parent and family functioning.

DETAILED DESCRIPTION:
There is considerable knowledge about how to help children with ABI during the first, acute and post-acute stages. Yet, impairments are often long lasting and, due to the vulnerability of children's developing brain, new problems may emerge or become increasingly problematic over time. Children with ABI may struggle at school and with peers, which can lead to or increase emotional difficulties, and reduce quality of life, affecting the children and their families. The local communities and the children's schools are, together with the families, often left responsible for dealing with the chronic challenges of pABI. Parents may experience considerable stress and develop emotional symptoms when a child suffers an ABI. As a result, the entire family may experience impaired functioning, which in turn may affect the long-term prognosis of the child with ABI.

Eighty families will be included in the study: 40 in the intervention group and 40 in the control group. The children will have a clinical ABI diagnosis, verified injury related intracranial abnormalities, and be at least one year post injury at inclusion. The children and/or their families must report enduring cognitive, emotional, social or physical challenges related to the brain injury. The intervention will be conducted in collaboration with the children's families, schools and their local health care providers. It consists of individualized goal-oriented strategies adapted to the home- and school-setting. Goal attainment scaling will be applied. In addition, psychoeducation will be provided to the family and school/local care providers on topics related to the child's injury. A parent group session will be held for discussions and knowledge transfer concerning family challenges after pABI, such as communication skills and parenting. The intervention will include 7 individualized meetings with the family (7 sessions whereof most will be videoconferences, but with the possibility of 1-2 of the sessions being home visits), one parent group seminar and 4 sessions with school and local health care providers during a period of 4-5 months.

Assessments will be conducted at baseline (T1), at the end of the intervention (T2, 4-5 months after inclusion) and one year after inclusion (T3). Baseline assessment includes a brief neuropsychological assessment of the children in addition to the outcome measures at T2 and T3. Outcome assessors will ble blinded to group allocation. Primary outcomes are change in parent-reported brain injury symptoms of the children and change in parenting self-efficacy. Secondary outcomes include change in child-rated severity of brain injury symptoms, change in unmet healthcare needs of the family, change in children's executive functioning in the home and school environment as assessed by parents, children and teachers, change in children's quality of life assessed by parents and children, change in family functioning, change in caregiver emotional symptoms, an evaluation of the intervention completed by parents, children and teachers in the intervention group, change in the perceived severity of the individually defined target outcome areas completed by children and parents, and change in goal attainment scaling in the intervention group.

The findings of this study will contribute to enhanced clinical expertise within pABI-rehabilitation on a specialist health care level, and will also be relevant for a wide array of health care professionals in the community as well as the educational system and parents of children with ABI.

ELIGIBILITY:
Inclusion Criteria:

* School-aged (6-16 years) children with clinical ABI-diagnosis and CT/MRI verified injury-related intracranial abnormalities, 1 year or more after injury. We anticipate including patients with the following etiologies: Traumatic brain injury (TBI), cerebrovascular incidents, anoxia, encephalitis and non-progressive brain tumors.
* The above-mentioned children, and/or their parents, report ABI-related cognitive, emotional, or behavioral problems that affect participation in activities with family, friends, school and/or community.
* The children attend school regularly, with or without injury-related adaptations.
* The family is able to actively participate in a goal-oriented approach, this includes speaking sufficiently Norwegian. An exception can be made for parents who speak English but are able to understand and read Norwegian.

Exclusion criteria:

* Patients with severe pre- or comorbid neurological or neuropsychiatric disorders that would confound assessment and/or treatment outcomes.
* Patients with brain tumors in active treatment or at great risk of relapse (i.e., unstable condition).
* Patients with severe psychiatric illness or children with injuries so severe that they are in institutionalized care most of the time.
* Parental severe psychiatric illness, drug abuse or indications of a history of or risk of domestic violence.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Change in parent-reported severity of children's brain injury symptoms | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the Health and Behavior Inventory (HBI) on a scale from 0 (Never) to 3 (Often), where higher score indicates more severe symptoms.
Change in parenting self-efficacy assessed with the assessment tool "Parenting Self-Efficacy (TOPSE)" | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  The Tool to measure Parenting Self-Efficacy (TOPSE) is rated on a scale from 0 (completely disagree) to 10 (completely agree). Higher total score on the questionnaire indicates higher parenting self-efficacy.

SECONDARY OUTCOMES:
Change in child-reported severity of brain injury symptoms | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the Health and Behavior Inventory (HBI) on a scale from 0 (Never) to 3 (Often), where higher score indicates more severe symptoms.
Change in unmet healthcare needs of the family | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the Family Needs Questionnaire - Pediatric version - FNQ-P on a scale from 1 (the need is not at all met) to 5 (completely met). Higher total score indicates higher level of met needs.
Change in children's executive functioning in the home and school environment | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the Behavior Rating Inventory of Executive Function 2 - BRIEF-2 on a 3-point scale: Never a problem, sometimes a problem or often a problem. Higher scaled score indicates higher level of problems with executive functioning.
Change in the children's quality of life | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the Pediatric Quality of Life Inventory - Peds-QL scored on a scale from 0 (never a problem) to 4 (almost always a problem). Higher scaled score indicates higher quality of life.
Change in family functioning | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the family Assessment Device - FAD on a 4-point scale: Strongly agree, agree, disagree and strongly disagree. Lower total scaled score represents better family functioning.
Change in depressive symptoms of the parents | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Assessed with the Patient Health Questionnaire 9 - PHQ-9 on a scale from 0 (not at all) to 3 (almost every day). Higher mean score reflects a higher level of depressive symptoms.
Change in anxiety symptoms of the parents | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Generalized Anxiety Disorder 7 - GAD-7 on a scale from from 0 (not at all) to 3 (almost every day). Higher mean score reflects a higher level of anxiety symptoms.
Evaluation of the intervention | Immediately after the intervention period (T2) (4-5 months after baseline)
  A custom-made evaluation questionnaire for the CICI Study will be completed by parents, children and teachers in the intervention group, as well as therapists. The Evaluation form is rated on a 5-point scale from "completely disagree" to "completely agree". Higher scaled score indicates higher degree of satisfaction.
Changes in the difficulty score (scale from 0 to 4) of the self- and parental perceived severity of the individually defined target outcome areas | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Each of the participating family members (parent(s) and child) nominate their three most important problems (target outcome areas) and how difficult they find them on a scale from 0 (not at all difficult) to 4 (very difficult), where . changes in the difficulty scores are evaluated. A negative change indicates a decrease in perceived difficulty.
Change in goal attainment scaling (GAS) in the CICI group | Change from baseline (T1) to immediately after the intervention period (T2) and one year after baseline (T3)
  Goal Attainment Scaling (GAS) is assessed by GAS-scaling of individually defined goals (scale from 1 to 5). A higher positive change reflects higher level of goal attainment.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Løvstad, PhD, Principal Investigator — Sunnaas Rehabilitation Hospital and University of Oslo
Locations (1):
- Sunnaas Rehabilitaion Hospital, Nesoddtangen, Akershus, Norway

REFERENCES:
- [Derived] Holthe IL, Rohrer-Baumgartner NM, Svendsen EJ, Roe C, Borgen IMH, Hauger SL, Ponsford JL, Egeland J, Wade S, Lovstad M. SMART-goal domains and goal attainment in an individualized, goal-oriented intervention for children with acquired brain injury and their families. Neuropsychol Rehabil. 2025 Jul;35(6):1229-1253. doi: 10.1080/09602011.2024.2402095. Epub 2024 Sep 16. PMID 39283234
- [Derived] Rohrer-Baumgartner N, Holthe IL, Svendsen EJ, Roe C, Egeland J, Borgen IMH, Hauger SL, Forslund MV, Brunborg C, Ora HP, Dahl HM, Bragstad LK, Killi EM, Sandhaug M, Kleffelgard I, Strand-Saugnes AP, Dahl-Hilstad I, Ponsford J, Winter L, Wade S, Lovstad M. Rehabilitation for children with chronic acquired brain injury in the Child in Context Intervention (CICI) study: study protocol for a randomized controlled trial. Trials. 2022 Feb 22;23(1):169. doi: 10.1186/s13063-022-06048-8. PMID 35193666